CLINICAL TRIAL: NCT03055624
Title: Prostate Artery Embolization for the Treatment of Symptomatic Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Andrew Picel, MD, Assistant Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161719
Record Dates: First submitted 2017-02-09; First posted 2017-02-16 (Actual); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Prostatic Hyperplasia, Benign; Enlarged Prostate With Lower Urinary Tract Symptoms
Keywords: prostate artery embolization (PAE); benign prostatic hyperplasia (BPH); lower urinary tract symptoms (LUTS)
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prostate artery embolization (Experimental): Single arm study of patients undergoing the prostate artery embolization procedure with Embosphere particles.
  Interventions: Device: Embosphere microparticles for prostate artery embolization

INTERVENTIONS:
Device: Embosphere microparticles for prostate artery embolization — Pelvic angiograms will be performed and microspheres delivered to the arteries supplying the prostate to alleviate symptoms of benign prostatic hyperplasia.

SUMMARY:
Investigator-initiated study to evaluate the safety and efficacy of prostate artery embolization for the treatment lower urinary tract symptoms in patients with benign prostatic hyperplasia

DETAILED DESCRIPTION:
This is a phase I/II, single center, prospective, single arm, investigational study to evaluate the safety and efficacy of prostate artery embolization (PAE) for treatment of severe lower urinary tract symptoms (LUTS) related to benign prostatic hyperplasia (BPH) in patients that have either failed or are intolerant to medical management. Once eligibility is confirmed, patients will undergo PAE with Embosphere Microspheres. Embolization will consist of a minimally invasive angiogram and treatment of the prostate arteries with the Embosphere particles to reduce blood flow to the prostate. Following treatment, patients will return for follow-up visits at 1, 6, 12, and 24 months post PAE.

ELIGIBILITY:
Inclusion Criteria:

1. Prostate volume between 40 and 300 cm3
2. Diagnosis of BPH with moderate to severe lower urinary tract symptoms (LUTS) defined as at least one of the following:

   * a. IPSS greater than 18
   * b. IPSS Quality of Life (QoL) assessment greater than 3
   * c. Qmax less than 12 mL/sec
3. Refractory or intolerant to medical management
4. Ineligibility for or refusal of surgical management
5. One of the following criteria:

   * a. Baseline prostate specific antigen (PSA) ≤2.5 ng/mL
   * b. Baseline PSA >2.5 ng/mL and ≤10 ng/mL AND free PSA ≥25% of total PSA
   * c. Baseline PSA >2.5 ng/mL and ≤10 ng/mL AND free PSA <25% of total PSA AND negative 12 core prostate biopsy in the past 12 months
   * d. Baseline PSA >10 ng/mL AND negative 12 core biopsy within the past 12 months.

Exclusion Criteria:

1. History of prostate, bladder or rectal malignancy. Biopsy proven urethral cancer.
2. History of rectal disease
3. Neurogenic bladder disorder due to multiple sclerosis, Parkinson's disease, spinal cord injury, diabetes, etc., as demonstrated on urodynamic testing.
4. Detrusor muscle failure, urethral stenosis, or urinary obstruction due to causes other than BPH, as demonstrated on urodynamic testing
5. Bladder diverticula greater than 5 cm or bladder stones greater than 2 cm
6. Cystolithiasis within the past three months
7. Baseline serum creatinine greater than 1.8
8. Evidence of tortuous or atherosclerotic blood vessels
9. Presence of collateral vessel pathways potentially endangering normal territories during embolization that cannot be bypassed with the microcatheter
10. Active urinary tract infection, interstitial cystitis, or prostatitis within the last 5 years
11. Coagulation disturbances not normalized by medical treatment
12. Allergy to iodinated contrast agents not responsive to steroid premedication regimen
13. Previous radical pelvic or rectal surgery, or pelvic irradiation
14. Prior surgical prostate intervention
15. Treatment with beta-blocker, antihistamine, anticonvulsant, or antispasmodic medication within 1 week of treatment UNLESS there has been a stable voiding pattern while medicated with the drug(s) for 6 months
16. Use of prostate active medications, including alpha blockers, anti-cholinergics, androgens, anti-androgens, gonadotropins-releasing hormonal analogs, PDE5-inhibitors, 5-alpha reductase inhibitors within 2 months of intervention, unless the medication is necessary to avoid symptom exacerbation and disability, in this case medication should not be initiated or dose adjusted within 1 month of study enrollment and dose should not be adjusted during the study period
17. Interest in future fertility
18. Mental condition or disorder that interferes with participants' ability to provide written informed consent
19. Current severe or uncontrolled disease (metabolic, hematologic, renal, hepatic, pulmonary, neurologic, cardiac, infectious or gastrointestinal) that in the Investigator's judgment makes the patient unsuitable for trial inclusion due to increased risk of complications
20. Known immunosuppression
21. Life expectancy less than 6 months

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Picel, MD, Principal Investigator — UCSD Medical Center
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were recruited in Interventional Radiology clinic from April 2017 to August 2018.
Pre-assignment Details: All patients enrolled were treated in the single treatment arm.
Period: Overall Study
Arm/Group | Prostate Artery Embolization
Started (9 patients enrolled in the study and underwent the PAE procedure.) | 9
Completed (The device received FDA IDE approval during the study. The study was closed at that time.) | 0
Not Completed | 9
Not completed — Study closed | 9

BASELINE CHARACTERISTICS:
Population: 9 patients enrolled and treated
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The study protocol was terminated before completion as the device was FDA approved and determined to be safe for the treated patient population.
Time Frame: 12 months
Population: Patients were assessed for adverse events during the time period the study was open
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 9
Participants | 3

2. Secondary Outcome: Change in International Prostate Symptom Score (IPSS)
Description: International Prostate Symptom Score change from baseline measured at 1 and 6 months. The IPSS scale grades lower urinary tract symptoms on a scale ranging from 0 (no symptoms) to 35 (severe). Patients answer 7 questions about symptoms they have had in the past month and grade each symptom severity for each question on a scale from 0 (not at all) to 5 (almost always). Change is reported as outcome measure time point minus baseline. A positive value indicates improved symptoms and negative value worsened symptoms.
Time Frame: baseline, 1 month, 6 month
Population: Data was not available for 1 participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 8
score on a scale
  1 month change | 16.1 (4.6)
  6 month change | 18.8 (4.6)

3. Secondary Outcome: Change in Post-void Residual (PVR) on Ultrasound
Description: PVR (mL) change from baseline measured at 1 and 6 months. Change is reported as outcome measure time point minus baseline. A negative value indicates less post-void residual and a positive value indicates greater PVR at each outcome time point.
Time Frame: baseline, 1 month, 6 month
Population: Data was not available for 4 participants.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 5
mL
  1 month change | -32 (66.5)
  6 month change | -84.8 (53.5)

4. Secondary Outcome: Change in Peak Urinary Flow Rate (Qmax)
Description: Change in Qmax measured at 1 and 6 months. Change is reported as outcome measure time point minus baseline. A positive value indicates improved Qmax and negative value indicates decreased Qmax at each outcome time point.
Time Frame: Baseline, 1 month, 6 month
Population: Data was not available for 4 participants
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 5
mL/sec
  1 month change | 2.4 (3.5)
  6 month change | 6 (6.1)

5. Secondary Outcome: Change in International Index of Erectile Dysfunction (IIEF)
Description: IIEF score change from baseline measured at 1 and 6 months. International Index of Erectile Function (IIEF) is a scale grading erectile function based on 5 questions. Questions are answered from 1 (low function) to 5 (high function). Total scores range from 5 to 25. A total score of 5-7 is severe erectile dysfunction, 8 to 11 is moderate erectile dysfunction, 12 to 16 is mild to moderate erectile dysfunction, 17 to 21 is mild erectile dysfunction, and 22-25 is no erectile dysfunction. Change is reported as outcome measure time point minus baseline. A positive value indicates improved erectile function and a negative indicates worsened erectile function.
Time Frame: baseline, 1 month, 6 month
Population: Data was not available for 5 participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 4
units on a scale
  1 month change | -1.3 (4.7)
  6 month change | 3 (2.8)

6. Secondary Outcome: Change in Prostate Volume (PV)
Description: Change in prostate volume measured at 1 and 6 months. Change is reported as outcome measure time point minus baseline. A negative value indicates decreased prostate volume and a positive value indicates increased prostate volume.
Time Frame: baseline, 1 month, 6 month
Population: Data was not available for 4 participants
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 5
mL
  1 month change | -30.7 (24.1)
  6 month change | -7.5 (13.1)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through the study period. 1 year data was available for the initial treated patients.
Description: Standard definitions used for adverse event and/or serious adverse event.
Arm/Group | Prostate Artery Embolization
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prostate Artery Embolization (N=9)
dysuria (Injury, poisoning and procedural complications) | 1 (1) — Patient experienced painful urination 1.5 days after the procedure. Symptom resolved without treatment.
Urinary retention (Renal and urinary disorders) | 1 (1) — Patient experienced urinary retention after the procedure requiring temporary catheter placement.
Skin wound (Renal and urinary disorders) | 1 (1) — Patient experienced a penile skin wound after treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT03055624/Prot_SAP_000.pdf